CLINICAL TRIAL: NCT07260006
Title: A Study on the Treatment Efficacy of Regimens With and Without Bismuth in Children With Helicobacter Pylori-Associated Peptic Ulcer Disease
Brief Title: Treatment Efficacy of Regimens With and Without Bismuth in Children With Helicobacter Pylori-Associated Peptic Ulcer Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Can Tho University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Mai Thùy Trang, Doctor, Can Tho University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2317/QD-DHYDCT
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-07

CONDITIONS: Helicobacter Pylori Infection; Peptic Ulcer
MeSH Terms: conditions — Peptic Ulcer | interventions — Amoxicillin; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bismuth quadruple therapy (Experimental): Patients in this arm will receive PPI, Amoxicillin, Metronidazole, and Bismuth for 14 days, with doses adjusted according to weight and age.
  Interventions: Drug: Bismuth quadruple therapy
- Triple therapy with PPI + Amoxicillin + Metronidazole (Experimental): Patients in this arm will receive PPI, Amoxicillin, Metronidazole for 14 days, with doses adjusted according to weight and age.
  Interventions: Drug: Triple therapy with PPI + Amoxicillin + Metronidazole

INTERVENTIONS:
Drug: Bismuth quadruple therapy — A 14-day regimen including proton pump inhibitor (PPI; esomeprazole [Nexium MUPS]), bismuth subcitrate (or bismuth subsalicylate), amoxicillin, and metronidazole. All drug doses are adjusted according to the participant's age and weight.
  Arms: Bismuth quadruple therapy
Drug: Triple therapy with PPI + Amoxicillin + Metronidazole — A 14-day regimen including proton pump inhibitor (PPI; esomeprazole [Nexium MUPS]), amoxicillin, and metronidazole.
  All drug doses are adjusted according to the participant's age and weight.
  Arms: Triple therapy with PPI + Amoxicillin + Metronidazole

SUMMARY:
The goal of this clinical trial is to learn if including bismuth in the treatment helps heal stomach and duodenal ulcers caused by Helicobacter pylori (H. pylori) in children.

The main questions it aims to answer are:

* Does a treatment plan with bismuth work better than a plan without bismuth to clear the infection?
* Is the bismuth plan more cost-effective while still safe and effective?

Researchers will compare two treatment groups to see which works better. Participants will:

* Take one of the two assigned treatment plans (with or without bismuth) for the standard treatment duration
* Visit the clinic for checkups and tests to confirm infection clearance and monitor side effects
* Keep a diary of symptoms, medication use, and any side effects

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with gastritis or peptic ulcer disease by upper gastrointestinal endoscopy or histopathology.
* Meets diagnostic criteria for Helicobacter pylori infection.
* Parent or legal guardian provides consent for the child to participate in the study.

Exclusion Criteria:

* Allergic to any of the medications in the treatment regimen.
* Use of antibiotics or bismuth within the past 4 weeks, or use of antacids, H2-receptor antagonists, or proton pump inhibitors within the past 2 weeks.
* Failure to return for follow-up visits after treatment.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Eradication rate of Helicobacter pylori infection between the two treatment regimens | Two weeks after discontinuation of acid suppression therapy following completion of the eradication regimen.
  The efficacy of the two regimens will be evaluated by comparing H. pylori eradication rates. Clinical examination and a urea breath test or stool antigen test will be performed after completion of therapy to confirm eradication. Patients will receive a 14-day treatment regimen, followed by an additional 2-4 weeks of proton pump inhibitor (PPI) therapy to promote healing of gastric or duodenal lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Can Tho Children's Hospital, Can Tho, Vietnam